CLINICAL TRIAL: NCT02160483
Title: Functional Brain Imaging and Psychological Testing in Women With Chronic Pelvic Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study is not feasible to conduct as functional brain imaging capability is inadequate. CIRB acknowledged in June 2016.
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013/728/D
Record Dates: First submitted 2014-05-25; First posted 2014-06-10 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Pelvis Pain Chronic; Endometriosis of Uterus
Keywords: Chronic pelvic pain; Endometriosis
MeSH Terms: conditions — Adenomyosis; Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Magnetic resonance imaging (Experimental): Functional magnetic resonance imaging using arterial spin labelling, functional connectivity, diffusion tensor imaging, magnetic resonance spectroscopy to evaluate women with chronic pelvic pain and/ or endometriosis
  Interventions: Other: Functional magnetic resonance imaging

INTERVENTIONS:
Other: Functional magnetic resonance imaging — 3 Tesla magnetic resonance imaging
  Other Names: FMRI

SUMMARY:
Functional magnetic resonance imaging in women with chronic pelvic pain using arterial spin labelling, functional connectivity, diffusion tensor imaging and magnetic resonance spectroscopy.

DETAILED DESCRIPTION:
Multimodal magnetic resonance neuroimaging will be utilised. Arterial spin labelling is tightly coupled with cerebral metabolism and can be used as a marker of neural activity. Resting state magnetic resonance imaging which measures synchronous activity across the brain, allows detection of functional connectivity of intrinsic brain network. Diffusion tensor imaging detects the anisotropic water diffusion in axonal fibres can provide information on connectivity and fibre tracts. Magnetic resonance spectroscopy would enable the levels of neurotransmitter to be elucidated.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pelvic pain
* Endometriosis

Exclusion Criteria:

* Contraindication to magnetic resonance imaging

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06 (Estimated); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with increase in insula anterior cingulate cortex signal on magnetic resonance imaging | 1 hour
  Magnetic resonance imaging using arterial spin labelling, functional connectivity, diffusion tensor imaging, magnetic resonance imaging

SECONDARY OUTCOMES:
Number of subjects in psychological testing with increased anxiety, depression and pain catastrophizing scores | 1 hour
  Anxiety, depression and pain catastrophizing scales used for psychological testing

CONTACTS AND LOCATIONS:
Overall Officials: Ban L Sng, FANZCA, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore